CLINICAL TRIAL: NCT06519279
Title: An International Multimodal Protocol for Assessing Freezing of Gait in Individuals Living with Parkinson's Disease
Brief Title: Freezing of Gait - Clinical Outcomes Assessment
Acronym: FOG-COA
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: KU Leuven (Other); Oregon Health and Science University (Other); University of Sydney (Other); Radbound University Medical Center (Unknown); University of Waterloo (Other); Emory University (Other); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 0608-23-TLV
Record Dates: First submitted 2024-07-03; First posted 2024-07-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: PD - Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Freezing Of Gait Patients: 15 patients with Parkinson disease with freezing of gait (group) in ON & OFF states
  Interventions: Device: Opals; Device: Axivity
- Non Freezing Of Gait Patients: 5 patients with Parkinson disease without freezing of gait (cohort) in ON & OFF states
  Interventions: Device: Opals; Device: Axivity

INTERVENTIONS:
Device: Opals — Five Oplas sensors were strategically placed on participants: one on each shin, one on each foot, and one on the lower back.
Device: Axivity — At the end of the first session, participants with FOG, will be fitted with an Axivity monitor. This is wearable sensor that will be attached to the participant's lower back (lumbar vertebrae 4-5) with hypoallergic medical tape by the researcher, and will be worn continuously for seven days.
  The Axivity monitor is a small (23 x 32.5 x 8.9 mm) and lightweight (11g) device that measures mobility via a tri-axial accelerometer and gyroscope and stores this data onboard, no GPS or other localization options are possible with this monitor. Participants will be given following guidelines concerning the use:
  The sensor is to be worn continuously during the seven-day period, i.e. also while sleeping and showering.
  The sensor is waterproof and can be worn during showering.

SUMMARY:
To develop a reliable and accurate clinician-reported outcome (ClinRO) measure (against a new and precise definition) and patient reported outcome (PRO) for use by clinicians and researchers to quantify the severity of Freezing of Gait (FOG).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease (PD) made by a neurologist according to the Movement Disorders Society guidelines;
2. Able to walk independently for a distance of 10 meters, without walking aid;
3. Absence of a Deep Brain Stimulator;
4. Stable PD treatment in the 4 weeks prior to participation that is not expected to change in the course of the study.
5. For patients with FOG: a score of ≥ 1 on the New Freezing Of Gait Questionnaire (NFOG-Q).

Exclusion Criteria:

1. Occurrence of any of the following within 3 months prior to informed consent: myocardial infarction, hospitalization for unstable angina, stroke, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), implantation of a cardiac resynchronization therapy device (CRTD), active treatment for cancer or other malignant disease, uncontrolled congestive heart disease (NYHA class >3), acute psychosis or major psychiatric disorders or continued substance abuse, other neurological (than PD) or orthopaedic impairment that significantly impacts on gait.
2. Unwilling to temporarily delay the morning anti-Parkinsonian medication.
3. Preganacy and

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FOG & NON-DOG
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Validate the newly-developed ClinRO | 12/2025
  Rate scale of freezing of gait to detect meaningful improvement in freezing of gait. The scale name is " Freezing Of Gait Severity Score". it consist a 8 trials, each one can be rate between 0 to 8. the scale consist a part of frequency of the freezing and part of cumulative duration. The higher the score, the more severe the stagnation and the lower it is, the less stagnation is present.

SECONDARY OUTCOMES:
Asses the importance of the FOG symptom for patients | 12/2025
  Severity of freezing of gait (FOG) symptoms and patient-reported impact on quality of life. The scale name is " Freezing Of Gait Severity Score". it consist a 8 trials, each one can be rate between 0 to 8. the scale consist a part of frequency of the freezing and part of cumulative duration. The higher the score, the more severe the stagnation and the lower it is, the less stagnation is present.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Saurasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided